CLINICAL TRIAL: NCT00537394
Title: The Optimized Treatment That Includes or Omits NRTIs Trial: A Randomized Strategy Study for HIV-1-Infected Treatment-Experienced Subjects Using the cPSS to Select an Effective Regimen
Brief Title: Optimizing Treatment for Treatment-Experienced, HIV-Infected People
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A5241; 10395 (Registry Identifier: DAIDS ES); ACTG A5241; OPTIONS
Expanded Access: Available
Record Dates: First submitted 2007-09-27; First posted 2007-10-01 (Estimated); Results first posted 2014-08-07 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2016-05

CONDITIONS: HIV Infections
Keywords: Treatment Experienced
MeSH Terms: conditions — HIV Infections | interventions — Enfuvirtide; Raltegravir Potassium; Darunavir; tipranavir; etravirine; Maraviroc

ARMS (3):
- A (Experimental): Regimen with higher predicted activity assigned by the study plus at least 2 NRTIs (personalized choice from expert recommendation) for 96 weeks. A 3-4 drug regimen was selected from the drugs listed to the right.
  Interventions: Drug: Enfuvirtide; Drug: Raltegravir; Drug: Darunavir; Drug: Tipranavir; Drug: Etravirine; Drug: Maraviroc
- B (Experimental): Regimen with higher predicted activity assigned by the study without NRTIs for 96 weeks. A 3-4 drug regimen was selected from the drugs listed to the right.
  Interventions: Drug: Enfuvirtide; Drug: Raltegravir; Drug: Darunavir; Drug: Tipranavir; Drug: Etravirine; Drug: Maraviroc
- C (Other): Regimen with lower predicted activity assigned plus at least 2 NRTIs (personalized choice from expert recommendation) for 96 weeks. A 3-4 drug regimen was selected from the drugs listed to the right.
  Interventions: Drug: Enfuvirtide; Drug: Raltegravir; Drug: Darunavir; Drug: Tipranavir; Drug: Etravirine; Drug: Maraviroc

INTERVENTIONS:
Drug: Enfuvirtide — 90mg subcutaneously twice daily
Drug: Raltegravir — 400 mg twice daily
Drug: Darunavir — Two 300-mg tablets twice daily, given with ritonavir 100mg twice daily (ritonavir not provided by the study)
Drug: Tipranavir — Two 250-mg capsules twice daily, given with ritonavir 100mg twice daily (ritonavir not provided by the study)
Drug: Etravirine — Two 100-mg tablets twice daily
Drug: Maraviroc — Dosage dependent on regimen in which maraviroc is included

SUMMARY:
The goal of anti-HIV therapy is to prevent HIV from replicating. Long-term control of HIV requires at least two anti-HIV drugs that are active against the virus. Drug resistance is a problem for many treatment-experienced, HIV-infected people. The purpose of this study was to determine the benefit of adding a nucleoside reverse transcriptase inhibitor (NRTI) to a new anti-HIV drug regimen for the suppression of HIV.

DETAILED DESCRIPTION:
Two or more fully active antiretrovirals (ARVs) are recommended for successful suppression of HIV. In people infected with resistant HIV virus, finding two drugs that are fully active against HIV can be a challenge. However, the new generation of anti-HIV drugs has been designed to suppress drug-resistant HIV. These drugs include the FDA-approved protease inhibitors (PIs) darunavir and tipranavir, the investigational non-nucleoside transcriptase inhibitor (nNRTI) etravirine, the FDA-approved fusion inhibitor enfuvirtide, the recently FDA-approved CCR5 inhibitor maraviroc, and the investigational integrase inhibitor raltegravir. Also, it is not yet known whether multiple, partially-active drugs have the same rate of success in suppressing HIV. The purpose of this study was to use HIV resistance testing to predict the potency of a suggested ARV regimen using second generation ARVs and determine if the benefits of adding NRTIs to this new drug regimen outweigh the risks of drug toxicity and pill burden. All participants had treatment experience or resistance to NRTIs, nNRTIs, and PIs, and received novel agents.

An active screening period (after enrollment but before randomization or treatment dispensation), occurred for up to 75 days for all participants, and study participation lasted an additional 96 weeks for those who qualified for either randomization or assignment (i.e. not randomized), to the study intervention. During active screening, all participants remained on their current drug regimen. During screening, phenotypic and genotypic HIV resistance tests were performed on participants' blood samples, as well as a coreceptor tropism assay. Using this information and medication history, the study team determined the best new regimen options for each participant. Each clinician, along with the study participant, then chose a new regimen based on the recommendations of the study team and the participant's preference.

Evaluation for study outcomes began when participants started their new regimen as assigned by either randomization or determined assignment. Stratification between Arms A (Add NRTIs) and B (Omit NRTIs) or Arm C (Non-randomized to Add NRTIs) was based on predicted activity of the new regimen. Those assigned to a regimen with higher predicted activity were randomly assigned to Arm A (Add NRTIs) or B (Omit NRTIs); those assigned a regimen predicted to have lower activity were not randomized, but were assigned to Arm C (Add NRTIs).

Participants in Arms A and C were instructed to take their newly assigned study regimen plus at least 2 NRTIs (personalized from expert recommendation and choice by local provider and participant) for 96 weeks. Participants in Arm B were instructed to take their newly assigned study regimen with no NRTIs for 96 weeks. Participants in all arms who met the primary efficacy outcome of regimen failure remained in the study in order to be followed for important secondary outcomes.

All participants were scheduled to have 13 clinical visits, which included blood collection. At some visits, urine collection and quality of life and adherence questionnaires occurred. A neurocognitive assessment was performed for all participants at time of starting the new study regimen. Participants may also have consented to have cerebrospinal fluid collected via lumbar puncture following study treatment assignment and/or at Week 24. Those participants who consented to cerebrospinal fluid collection also had neurocognitive assessments at the times of collections. Participants were responsible for obtaining certain ARVs not provided by the study, including the ARVs they during the active screening period.

The primary and secondary study objectives and comparisons relate to the randomized arms, and therefore, results are not provided for the non-randomized arm (C). The purpose of the non-randomized arm (C) was to include persons higher baseline resistance (and thus, lower activity scores) in order to address an exploratory objective related to the predictive power of these activity scores (and thus a larger range of scores by inclusion of arm C), on certain, virologic outcomes.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection
* Triple-class drug experience or resistance. More information on this criterion can be found in the protocol.
* Currently on a failing PI-containing regimen that includes 2 other ARVs with no regimen change for 8 weeks prior to study screening
* HIV viral load of 1000 copies/ml or more
* Hepatitis B surface antigen negative within 90 days of study entry
* Able to obtain NRTIs and ritonavir and have required ARVs at time of starting study intervention
* Willing to use acceptable forms of contraception
* Parent or legal guardian willing to provide consent, if applicable
* CD4 count result from a specimen drawn within 120 days prior to study entry
* If any previous HIV-1 viral co-receptor tropism result is available, then most recent specimen date and the tropism result of that specimen AND specimen date and tropism result of any test with either X4 or D/M result, if different from the first specimen, must be available

Inclusion Criteria continued:

* Receipt of successful phenotype/genotype resistance results within 105 days prior to study treatment intervention assignment
* Study team identification of a study regimen and at least 2 NRTIs for participant to take
* Certain abnormal laboratory values. More information on this criterion can be found in the protocol.

Exclusion Criteria:

* Chronic, active hepatitis B virus infection (hepatitis B surface antigen positive or HBV DNA positive)
* Taking certain medications. More information on this criterion can be found in the protocol.
* Known allergy/sensitivity to components of two or more of the study-provided drugs or their formulations. For maraviroc, this includes hypersensitivity or history of allergy to soy lecithin or peanuts.
* Active drug or alcohol use that, in the opinion of the investigator, may interfere with the study
* Pregnancy or breastfeeding
* Use of any immunomodulator (interferons, interleukins, systemic corticosteroids, or cyclosporine), vaccine, or investigational therapy within 30 days prior to study treatment allocation/assignment
* Require certain medications prohibited with study treatment
* Serious illness requiring systemic treatment or hospitalization. Participants who complete therapy or are clinically stable on therapy for at least 14 days prior to study treatment allocation are not excluded.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 517 (Actual)
Dates: Start 2008-01; Primary Completion 2012-05 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen T. Tashima, MD, Study Chair — Brown University; Richard H. Haubrich, MD, Study Chair — Division of Infectious Diseases, UCSD Antiviral Research Center
Locations (64):
- United States (61):
  - Alabama Therapeutics CRS, Birmingham, Alabama
  - Miller Children's Hosp. Long Beach CA NICHD CRS, Long Beach, California
  - University of Southern California CRS, Los Angeles, California
  - Usc La Nichd Crs, Los Angeles, California
  - UCLA CARE Center CRS, Los Angeles, California
  - UCLA-Los Angeles/Brazil AIDS Consortium (LABAC) CRS, Los Angeles, California
  - Stanford AIDS Clinical Trials Unit CRS, Palo Alto, California
  - UCSD Antiviral Research Center CRS, San Diego, California
  - Ucsf Hiv/Aids Crs, San Francisco, California
  - Univ. of California San Francisco NICHD CRS, San Francisco, California
  - University of Colorado Hospital CRS, Aurora, Colorado
  - Denver Public Health CRS, Denver, Colorado
  - Georgetown University CRS (GU CRS), Washington D.C., District of Columbia
  - Children's National Med. Ctr. ATN CRS, Washington D.C., District of Columbia
  - Howard Univ. Washington DC NICHD CRS, Washington D.C., District of Columbia
  - Pediatric Perinatal HIV Clinical Trials Unit CRS, Miami, Florida
  - The Ponce de Leon Center CRS, Atlanta, Georgia
  - Northwestern University CRS, Chicago, Illinois
  - Rush University CRS, Chicago, Illinois
  - Tulane Univ. New Orleans NICHD CRS, New Orleans, Louisiana
  - IHV Baltimore Treatment CRS, Baltimore, Maryland
  - Johns Hopkins University CRS, Baltimore, Maryland
  - Massachusetts General Hospital CRS (MGH CRS), Boston, Massachusetts
  - Brigham and Women's Hospital Therapeutics Clinical Research Site (BWH TCRS) CRS, Boston, Massachusetts
  - Bmc Actg Crs, Boston, Massachusetts
  - Boston Medical Center Ped. HIV Program NICHD CRS, Boston, Massachusetts
  - Beth Israel Deaconess Med. Ctr., ACTG CRS, Boston, Massachusetts
  - Wayne State Univ. CRS, Detroit, Michigan
  - Henry Ford Hosp. CRS, Detroit, Michigan
  - Washington University Therapeutics (WT) CRS, St Louis, Missouri
  - Cooper Univ. Hosp. CRS, Camden, New Jersey
  - New Jersey Medical School Clinical Research Center CRS, Newark, New Jersey
  - Rutgers - New Jersey Medical School CRS, Newark, New Jersey
  - Weill Cornell Chelsea CRS, New York, New York
  - NY Univ. HIV/AIDS CRS, New York, New York
  - Nyu Ny Nichd Crs, New York, New York
  - Metropolitan Hosp. NICHD CRS, New York, New York
  - Columbia P&S CRS, New York, New York
  - Columbia IMPAACT CRS, New York, New York
  - Harlem ACTG CRS, New York, New York
  - Trillium Health ACTG CRS, Rochester, New York
  - Univ. of Rochester ACTG CRS, Rochester, New York
  - Bronx-Lebanon Hosp. Ctr. CRS, The Bronx, New York
  - Chapel Hill CRS, Chapel Hill, North Carolina
  - Duke Univ. Med. Ctr. Adult CRS, Durham, North Carolina
  - Cincinnati CRS, Cincinnati, Ohio
  - Case Clinical Research Site, Cleveland, Ohio
  - MetroHealth CRS, Cleveland, Ohio
  - Ohio State University CRS, Columbus, Ohio
  - The Research & Education Group-Portland CRS, Portland, Oregon
  - Penn Therapeutics, CRS, Philadelphia, Pennsylvania
  - Thomas Jefferson Univ. Med. Ctr. CRS, Philadelphia, Pennsylvania
  - University of Pittsburgh CRS, Pittsburgh, Pennsylvania
  - The Miriam Hospital Clinical Research Site (TMH CRS) CRS, Providence, Rhode Island
  - St. Jude Children's Research Hospital CRS, Memphis, Tennessee
  - Vanderbilt Therapeutics (VT) CRS, Nashville, Tennessee
  - Trinity Health and Wellness Center CRS, Dallas, Texas
  - Houston AIDS Research Team CRS, Houston, Texas
  - Texas Children's Hospital CRS, Houston, Texas
  - Virginia Commonwealth Univ. Medical Ctr. CRS, Richmond, Virginia
  - University of Washington AIDS CRS, Seattle, Washington
- Puerto Rico (3):
  - Puerto Rico AIDS Clinical Trials Unit CRS, San Juan
  - University of Puerto Rico Pediatric HIV/AIDS Research Program CRS, San Juan
  - San Juan City Hosp. PR NICHD CRS, San Juan

REFERENCES:
- [Background] Altmann A, Beerenwinkel N, Sing T, Savenkov I, Doumer M, Kaiser R, Rhee SY, Fessel WJ, Shafer RW, Lengauer T. Improved prediction of response to antiretroviral combination therapy using the genetic barrier to drug resistance. Antivir Ther. 2007;12(2):169-78. doi: 10.1177/135965350701200202. PMID 17503659
- [Background] Eshleman SH, Husnik M, Hudelson S, Donnell D, Huang Y, Huang W, Hart S, Jackson B, Coates T, Chesney M, Koblin B. Antiretroviral drug resistance, HIV-1 tropism, and HIV-1 subtype among men who have sex with men with recent HIV-1 infection. AIDS. 2007 May 31;21(9):1165-74. doi: 10.1097/QAD.0b013e32810fd72e. PMID 17502727
- [Background] Geretti AM. Clinical implications of HIV drug resistance to nucleoside and nucleotide reverse transcriptase inhibitors. AIDS Rev. 2006 Oct-Dec;8(4):210-20. PMID 17219736
- [Background] Mallolas J, Blanco J, Labarga P, Vergara A, Ocampo A, Sarasa M, Arnedo M, Lopez-Pua Y, Garcia J, Juega J, Guelar A, Terron A, Dalmau D, Garcia I, Zarraga M, Martinez E, Carne X, Pumarola T, Escayola R, Gatell J. Inhibitory quotient as a prognostic factor of response to a salvage antiretroviral therapy containing ritonavir-boosted saquinavir. The CIVSA Study. HIV Med. 2007 May;8(4):226-33. doi: 10.1111/j.1468-1293.2007.00464.x. PMID 17461850
- [Derived] Gandhi RT, Tashima KT, Smeaton LM, Vu V, Ritz J, Andrade A, Eron JJ, Hogg E, Fichtenbaum CJ. Long-term Outcomes in a Large Randomized Trial of HIV-1 Salvage Therapy: 96-Week Results of AIDS Clinical Trials Group A5241 (OPTIONS). J Infect Dis. 2020 Apr 7;221(9):1407-1415. doi: 10.1093/infdis/jiz281. PMID 31135883
- [Derived] Tashima KT, Smeaton LM, Fichtenbaum CJ, Andrade A, Eron JJ, Gandhi RT, Johnson VA, Klingman KL, Ritz J, Hodder S, Santana JL, Wilkin T, Haubrich RH; A5241 Study Team. HIV Salvage Therapy Does Not Require Nucleoside Reverse Transcriptase Inhibitors: A Randomized, Controlled Trial. Ann Intern Med. 2015 Dec 15;163(12):908-17. doi: 10.7326/M15-0949. Epub 2015 Nov 24. PMID 26595748

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects recruited between February 2008 and May 2011 from participating ACTG, IMPAACT, and ATN network sites located in the continental US and Puerto Rico.
Pre-assignment Details: A total of 104 exclusions among 517 enrolled to active screening but prior to assignment and dispensation of study treatment were due to any of the following: no resistance/tropism test results, not willing to accept any ARV study regimens, changes to current PI based ARV regimen or non-adherence, or changes with respect to eligibility criteria.
Groups:
- Add NRTIs (Randomized) to Individualized Regimen (cPSS > 2.0): [Arm A]Individualized ARV study regimen with antiretroviral potency defined as continuous phenotype sensitivity score (cPSS) greater than 2.0 recommended and chosen prior to randomization. To this regimen, an individualized NRTI combination of at least 2 drugs from this class, chosen prior to randomization, was also started.
- Omit NRTIs (Randomized) From Individualized Regimen(cPSS > 2): [Arm B] Individualized ARV study regimen with antiretroviral potency defined as continuous phenotype sensitivity score (cPSS) greater than 2.0 recommended and chosen prior to randomization. To this regimen, an individualized NRTI combination of at least 2 drugs from this class, chosen prior to randomization, was omitted, and any NRTIs the participant had been taking prior to randomization were to be permanently discontinued.
- Non-randomized Group: Add NRTIs to Individual Regimen cPSS <=2: [Non-randomized Group C] : Among persons whose ARV resistance and history profile precluded any of the 20 possible ARV regimens having high enough potential potency (cPSS <=2), treatment was assigned rather than being a randomized. To their regimen, individualized NRTI combination of at least 2 drugs from this class were added in order to form the most potent ARV regimen possible.
Period: First Year of Follow-up
Arm/Group | Add NRTIs (Randomized) to Individualized Regimen (cPSS > 2.0) | Omit NRTIs (Randomized) From Individualized Regimen(cPSS > 2) | Non-randomized Group: Add NRTIs to Individual Regimen cPSS <=2
Started | 181 | 179 | 53
Completed | 169 (Completed refers to completing first 48 weeks of follow-up.) | 168 (Completed refers to completing first 48 weeks of follow-up.) | 50
Not Completed | 12 | 11 | 3
Not completed — Death | 7 | 0 | 0
Not completed — Severe debilitation | 1 | 0 | 1
Not completed — Withdrawal by Subject | 3 | 6 | 1
Not completed — Lost to Follow-up | 1 | 5 | 1
Period: 2nd Year of Follow-up
Arm/Group | Add NRTIs (Randomized) to Individualized Regimen (cPSS > 2.0) | Omit NRTIs (Randomized) From Individualized Regimen(cPSS > 2) | Non-randomized Group: Add NRTIs to Individual Regimen cPSS <=2
Started | 169 | 168 | 50
Completed | 158 | 159 | 44
Not Completed | 11 | 9 | 6
Not completed — Death | 4 | 1 | 2
Not completed — Withdrawal by Subject | 0 | 1 | 2
Not completed — Lost to Follow-up | 6 | 7 | 2
Not completed — Clinic site closure | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Everyone randomized (ITT study sample), plus non-randomized group.
Groups:
- Add NRTIs (Randomized) to Individualized Regimen (cPSS > 2.0): Individualized ARV study regimen with antiretroviral potency defined as continuous phenotype sensitivity score (cPSS) greater than 2.0 recommended and chosen prior to randomization. To this regimen, an individualized NRTI combination of at least 2 drugs from this class, chosen prior to randomization, was also started.
- Omit NRTIs (Randomized) From Individualized Regimen(cPSS > 2): Individualized ARV study regimen with antiretroviral potency defined as continuous phenotype sensitivity score (cPSS) greater than 2.0 recommended and chosen prior to randomization. To this regimen, an individualized NRTI combination of at least 2 drugs from this class, chosen prior to randomization, was omitted, and any NRTIs the participant had been taking prior to randomization were to be permanently discontinued.
- Non-randomized Group: Add NRTIs to Individual Regimen cPSS <=2: Among persons whose ARV resistance and history profile precluded any of the 20 possible ARV regimens having high enough potential potency (cPSS <=2), treatment was assigned rather than being a randomized. To their regimen, individualized NRTI combination of at least 2 drugs from this class were added in order to form the most potent ARV regimen possible.
- Total: Total of all reporting groups
Arm/Group | Add NRTIs (Randomized) to Individualized Regimen (cPSS > 2.0) | Omit NRTIs (Randomized) From Individualized Regimen(cPSS > 2) | Non-randomized Group: Add NRTIs to Individual Regimen cPSS <=2 | Total
Number analyzed (Participants) | 181 | 179 | 53 | 413
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6 | 8 | 3 | 17
  Between 18 and 65 years | 173 | 168 | 50 | 391
  >=65 years | 2 | 3 | 0 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.7 (10.8) | 44.1 (11.7) | 43.1 (10.7) | 44.3 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 47 | 6 | 99
  Male | 135 | 132 | 47 | 314
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 37 | 46 | 14 | 97
  Not Hispanic or Latino | 141 | 132 | 38 | 311
  Unknown or Not Reported | 3 | 1 | 1 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 2 | 1 | 6
  Asian | 0 | 4 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 81 | 72 | 20 | 173
  White | 88 | 87 | 29 | 204
  More than one race | 1 | 2 | 0 | 3
  Unknown or Not Reported | 8 | 11 | 2 | 21
Region of Enrollment [Number; unit: participants]
  United States | 181 | 179 | 53 | 413
CD4 count, continuous [Mean (Standard Deviation); unit: cells/mm^3] | 252.3 (194.9) | 245.6 (195.1) | 154.8 (170.1) | 236.9 (194.2)
Plasma HIV-1 RNA, continuous [Median (Inter-Quartile Range); unit: log10 copies/mL] | 4.2 [3.6 to 4.7] | 4.2 [3.6 to 4.6] | 4.4 [4.1 to 4.8] | 4.2 [3.6 to 4.6]

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants With Regimen Failure, Defined as a Confirmed Virologic Failure or Discontinuation of Randomized NRTI Component of Study Treatment
Description: Virologic failure defined as confirmed plasma HIV-1 RNA meeting 1 of the following 4 criteria: < 1.0 log10 copies/mL reduction from baseline level and >= 200 copies/mL at or after week 12 evaluation; >= 200 copies/mL after 1 measurement < 200 copies/mL; absence of any values < 200 copies/mL by and including week 24 evaluation; >= 200 copies/mL at week 48 evaluation. Discontinuation of Randomized NRTI component of Study Treatment is defined as permanently stopping all NRTIs among those randomized to add NRTIs, or starting any NRTI among those randomized to omit NRTIs. Subjects leaving the study for reasons other than death, relocation, incarceration, or site closure were reviewed for the discontinuation outcome by a blinded, independent panel. Additionally, any participant failing to start study treatment after randomization and prior to closure was also reviewed. Results report percent of participants reaching regimen failure outcome by week 48 evaluation using Kaplan-Meier method.
Time Frame: From study entry to end of Week 48 evaluation window
Population: Analysis uses intent to treat population, among the two randomized arms only.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Add NRTIs (Randomized) to Individualized Regimen (cPSS > 2.0) | Omit NRTIs (Randomized) From Individualized Regimen(cPSS > 2)
Number analyzed (Participants) | 181 | 179
percentage of participants | 26.0 [19.6 to 32.3] | 29.8 [23.1 to 36.6]
Statistical Analysis 1: Comparison: Add NRTIs (Randomized) to Individualized Regimen (cPSS > 2.0) vs Omit NRTIs (Randomized) From Individualized Regimen(cPSS > 2); Null Hypothesis was that omitting NRTIs is inferior to adding NRTIs for the outcome of regimen failure through 48 weeks; Test type: Non-Inferiority or Equivalence — Non-inferiority margin defined as 15 percentage points. If the confidence interval for the difference in regimen failure between omitting versus adding NRTIs was fully below 15 percentage points, then omitting NRTIs would be concluded to be not inferior to adding NRTIs for this outcome; Risk Difference (RD) = 3.2, 95% CI 2-sided [-6.1 to 12.5] — Endpoint rates with standard errors calculated from Kaplan-Meier curves for each treatment group and stratum. Differences in week 48 failure proportions by treatment calculated weighted by the inverse of the variance in each stratum

2. Secondary Outcome: Time From Treatment Dispensation to First Grade 3 or Higher (and at Least One Grade Higher Than Baseline) Signs/Symptom or Laboratory Abnormality
Description: Events following permanent discontinuation of NRTI assignment are excluded (i.e. censoring at time of this event, if applicable). Week 96 study visit could occur up to 110 weeks following randomization. Censoring time was the latest study visit when participant was evaluated or when NRTI assignment was discontinued (when applicable). Event time was the exact number of weeks following treatment initiation when the qualifying sign/symptom started (for those safety events triggered by a sign/symptom), or exact number of weeks following treatment initiation when specimen from qualifying laboratory result was drawn (for those safety events triggered by a laboratory abnormality).
Time Frame: From treatment dispensation to week 96 study visit
Population: Only randomized participants included. Persons not starting study treatment excluded.
Measure: Number (95% Confidence Interval); unit: weeks
Arm/Group | Add NRTIs (Randomized) to Individualized Regimen (cPSS > 2.0) | Omit NRTIs (Randomized) From Individualized Regimen(cPSS > 2)
Number analyzed (Participants) | 180 | 177
weeks
  5th percentile | 3.1 [1.9 to 4.6] | 3.9 [0.9 to 4.6]
  25th percentile | 24.7 [12.0 to 47.0] | 25.3 [24.0 to 35.9]
  50th percentile | NA [72.1 to NA] — Not estimable as the estimate and upper limit for survival function at all weeks is above 50% | 97.7 [63.0 to NA] — Not estimable as the upper limit for survival function at all weeks is above 50%

3. Secondary Outcome: Time From Treatment Dispensation to First Study ARV Modification (Excluding NRTIs, if Applicable)
Description: First study ARV modification included any discontinuation or substitution of any chosen and initiated ARV for any reason. Events prompting study medication change could include protocol required (e.g. safety), protocol recommended but not required (e.g. virologic failure), or participant motivated (such as non-adherence, loss to follow-up or death; in other words, not protocol recommended or required). Event times were the exact weeks from treatment initiation to the time of qualifying regimen modification. Censoring times were the exact weeks from treatment initiation to the last date of study drugs. The week 96 (final study visit) could occur up through 110 weeks following randomization.
Time Frame: From treatment dispensation to week 96 study visit
Population: Only randomized participants included, and those who never started study treatment were excluded.
Measure: Number (95% Confidence Interval); unit: weeks
Arm/Group | Add NRTIs (Randomized) to Individualized Regimen (cPSS > 2.0) | Omit NRTIs (Randomized) From Individualized Regimen(cPSS > 2)
Number analyzed (Participants) | 180 | 177
weeks
  5th percentile | 9.0 [1.1 to 29.7] | 24.0 [4.0 to 35.6]
  10th percentile | 31.1 [14.7 to 51.1] | 38.0 [24.4 to 67.7]
  25th percentile | 98.0 [82.7 to NA] — Not estimable as the upper limit for survival function at all weeks is above 75%. | NA [84.4 to NA] — Not estimable as the estimate for survival function at all weeks is above 75%.

4. Secondary Outcome: Time From Randomization to Discontinuation of Randomized NRTI Component of Study Treatment
Description: Discontinuation of Randomized NRTI component of Study Treatment is defined as permanently stopping all NRTIs among those randomized to add NRTIs, or starting any NRTI among those randomized to omit NRTIs. Subjects leaving the study for reasons other than death, relocation, incarceration, or site closure were reviewed for meeting this outcome by a blinded, independent panel. Additionally, any participant failing to start study treatment after randomization and prior to closure was also reviewed. Event times were scheduled study weeks when discontinuation events occurred. Censoring times were latest scheduled study visit weeks with evaluation.
Time Frame: From randomization to week 96 study visit
Population: All randomized participants included (i.e. ITT analysis).
Measure: Number (95% Confidence Interval); unit: weeks
Arm/Group | Add NRTIs (Randomized) to Individualized Regimen (cPSS > 2.0) | Omit NRTIs (Randomized) From Individualized Regimen(cPSS > 2)
Number analyzed (Participants) | 181 | 179
weeks
  1st percentile | 0 [0 to 1] | 0 [0 to 12]
  5th percentile | 36 [1 to NA] — Not estimable as the upper limit for survival function at all weeks is above 95%. | 36 [4 to 36]
  10th percentile | NA [36 to NA] — Not estimable as the estimate for survival function at all weeks is above 90%. | 48 [36 to 84]

5. Secondary Outcome: Time From Randomization to Confirmed Virological Failure
Description: Virologic failure defined as confirmed (two consecutive) plasma HIV-1 RNA meeting 1 of the following 4 criteria: < 1.0 log10 copies/mL reduction from baseline level and >= 200 copies/mL at or after week 12 evaluation; >= 200 copies/mL after 1 measurement < 200 copies/mL; absence of any values < 200 copies/mL by and including week 24 evaluation; >= 200 copies/mL at week 48 evaluation. Event time was the scheduled study visit week when the initial plasma HIV-1 RNA specimen meeting the failure definition was collected. Censoring time was the latest scheduled study visit week when a plasma HIV-1 RNA specimen was collected and tested.
Time Frame: From randomization to week 96 study visit
Population: ITT (all randomized participants) included.
Measure: Number (95% Confidence Interval); unit: weeks
Arm/Group | Add NRTIs (Randomized) to Individualized Regimen (cPSS > 2.0) | Omit NRTIs (Randomized) From Individualized Regimen(cPSS > 2)
Number analyzed (Participants) | 181 | 179
weeks
  5th percentile | 12 [8 to 12] | 12 [8 to 12]
  10th percentile | 12 [12 to 16] | 12 [12 to 16]
  25th percentile | 48 [24 to NA] — Not estimable as the upper limit for survival function at all weeks is above 75%. | 48 [36 to NA] — Not estimable as the upper limit for survival function at all weeks is above 75%.

6. Secondary Outcome: Number of Participants With Plasma HIV-1 Viral Load < 50 Copies/ml
Description: Number of participants with plasma HIV-1 Viral load < 50 copies/mL at study visit weeks 24, 48, and 96. Closest observed result between 20 and up to 30 weeks (for week 24), between 42 and up to 54 (for week 48), and between 90 and up to 110 (for week 96) used if multiple results available. Missing values excluded.
Time Frame: At Weeks 24, 48, 96
Population: ITT - among 2 randomized arms only; closest value to scheduled week used if multiple values available; missing values excluded. Numbers analyzed at each time point represent those with a valid RNA result.
Measure: Number; unit: participants
Arm/Group | Add NRTIs (Randomized) to Individualized Regimen (cPSS > 2.0) | Omit NRTIs (Randomized) From Individualized Regimen(cPSS > 2)
Number analyzed (Participants) | 181 | 179
participants
  Week 24: Number with RNA < 50 c/mL (N=170; N=171) | 122 | 117
  Week 48: Number with RNA < 50 c/mL (N=169; N=165) | 112 | 106
  Week 96: Number with RNA < 50 c/mL (N=158; N=158) | 107 | 109

7. Secondary Outcome: Change in Plasma HIV-1 Viral Load From Baseline to Week 1
Description: Method of Kaplan and Meier used to accommodate left-censoring for those whose week 1 levels < 50 copies/mL.
Time Frame: From baseline to Week 1 evaluation
Population: Modified intent to treat population among two randomized arms only: 2 participants (both in Omit NRTIs arm) were excluded because their baseline and week 1 RNA levels were both < 50 copies/mL.
Measure: Median (Inter-Quartile Range); unit: log10 copies/mL
Arm/Group | Add NRTIs (Randomized) to Individualized Regimen (cPSS > 2.0) | Omit NRTIs (Randomized) From Individualized Regimen(cPSS > 2)
Number analyzed (Participants) | 172 | 173
log10 copies/mL | 1.3 [0.9 to 1.6] | 1.4 [0.9 to 1.6]

8. Secondary Outcome: Change in Summarized Quality of Life Score
Description: Quality-of-life score at each evaluation based upon a single question assessing participants' self-report of general health with a range of 0 (representing worst health status) to 100 (representing perfect health).
Time Frame: At study entry and Weeks 24, 48, 96
Population: Two randomized arms only.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Add NRTIs (Randomized) to Individualized Regimen (cPSS > 2.0) | Omit NRTIs (Randomized) From Individualized Regimen(cPSS > 2)
Number analyzed (Participants) | 181 | 179
units on a scale
  Change from baseline to week 24 (N=165; N=165) | 0 [-5 to 15] | 5 [0 to 15]
  Change from baseline to week 48 (N=161; N=158) | 0 [-10 to 15] | 0 [-5 to 10]
  Change from baseline to week 96 (N=155; N=154) | 0 [-5 to 15] | 0.5 [-3 to 19]

9. Secondary Outcome: Number of Participants Self-reporting Non-adherence to Assigned Study ARVS (Excluding NRTIs, if Applicable)
Description: Results represent self-report of non-adherence during the 4-day period prior to the outcome evaluation visit. Participants in follow-up for whom these data are missing for any reason are inferred as not-adherent.
Time Frame: At Weeks 24 and 48
Population: Persons not starting study treatment, or not receiving assigned study treatment by randomization were excluded from all analyses. If person no longer in study follow-up before beginning of week 24 or 48 evaluation window, additionally excluded as applicable.
Measure: Number; unit: participants
Arm/Group | Add NRTIs (Randomized) to Individualized Regimen (cPSS > 2.0) | Omit NRTIs (Randomized) From Individualized Regimen(cPSS > 2)
Number analyzed (Participants) | 180 | 177
participants
  Week 24 (N=170; N=172) | 25 | 26
  Week 48 (N=167; N=163) | 30 | 26

10. Secondary Outcome: Change in Cardiovascular Risk Score From Baseline
Description: Cardiovascular risk score defined by Framingham providing an estimate of the probability of developing cardiovascular disease over the next 10-year period. Persons with a historical cardiovascular event (CAD, cerebro- or peripheral- vascular disorder, MI or stroke), were excluded, and scores were not calculated at follow-up times after individuals had a cardiovascular event. Missing values for input data (e.g. smoking status) resulted in a missing value for Framingham score.
Time Frame: At Weeks 24, 48, and 96
Population: Persons not starting treatment (N=1; N=2), who had cardiovascular disease prior to study entry (N=12; N=8), or were missing input values needed to calculate a baseline Framingham score (N= 6; N=4), were excluded.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Add NRTIs (Randomized) to Individualized Regimen (cPSS > 2.0) | Omit NRTIs (Randomized) From Individualized Regimen(cPSS > 2)
Number analyzed (Participants) | 162 | 165
units on a scale
  Week 24 (N= 150; N=147) | -0.7 (4.4) | 0.3 (4.9)
  Week 48 (N=143; N=144) | 0.1 (4.3) | 0.8 (4.9)
  Week 96 (N=129; N=132) | 0.5 (5.2) | 1.1 (5.0)

11. Secondary Outcome: Change in CD4 Count From Baseline
Description: Baseline CD4 calculated as average of pre-entry and entry values. Closest observed result between 42 and up to 54 weeks (for week 48) or between 90 and up to 110 weeks (for week 96), used if multiple results available. Missing values excluded.
Time Frame: From study entry to Weeks 48 and 96
Population: All subjects in the two randomized arms were assessed.
Measure: Median (Inter-Quartile Range); unit: cells/mm^3
Arm/Group | Add NRTIs (Randomized) to Individualized Regimen (cPSS > 2.0) | Omit NRTIs (Randomized) From Individualized Regimen(cPSS > 2)
Number analyzed (Participants) | 181 | 179
cells/mm^3
  Change from entry to week 48 (N=166; N=163) | 105.5 [46.0 to 214.0] | 89.5 [33.0 to 166.5]
  Change from entry to week 96 (N= 154; N=157) | 140.8 [39.0 to 244.5] | 115.5 [31.5 to 229.5]

12. Secondary Outcome: Time From Treatment Dispensation to Serious Non-AIDS-defining Events
Description: Serious Non-AIDS defining Events were adjudicated by independent and blinded review and possible events included serious diagnoses in the following disease areas: liver, cardiovascular, end-stage renal, non-AIDS malignancy, and diabetes mellitus. Week 96 study visit could take place up to 110 weeks following randomization. Event times were the exact weeks following treatment initiation corresponding to the diagnosis dates of the qualifying serious non-AIDS defining events. Censoring times were the weeks following treatment initiation corresponding to the latest study visit.
Time Frame: From treatment initiation to week 96 study visit
Population: Randomized participants were included, and those not starting study treatment were excluded.
Measure: Number (95% Confidence Interval); unit: weeks
Arm/Group | Add NRTIs (Randomized) to Individualized Regimen (cPSS > 2.0) | Omit NRTIs (Randomized) From Individualized Regimen(cPSS > 2)
Number analyzed (Participants) | 180 | 177
weeks
  1st percentile | 4.9 [1.9 to 26.0] | 29.3 [23.1 to 41.3]
  5th percentile | 60.0 [13.0 to NA] — Not estimable as the upper limit for survival function at all weeks are above 95%. | NA [31.7 to NA] — Not estimable as the estimates and upper limit for survival function at all weeks are above 95%.

13. Secondary Outcome: Number of Participants With Change in Virus Co-receptor Tropism Among Those With R5-only Tropic Virus at Study Entry
Description: HIV Co-receptor tropism test result of either dual/mixed or evidence of X4 using virus from sample collected at confirmed virologic failure.
Time Frame: From study entry to time of confirmed virological failure (up to 96 weeks)
Population: Only randomized participants with R5-tropic virus at study entry (N=89; N=88), and who experienced confirmed virologic failure (N=27; N=22) during follow-up, and who had a tropism test following failure are included.
Measure: Number; unit: participants
Arm/Group | Add NRTIs (Randomized) to Individualized Regimen (cPSS > 2.0) | Omit NRTIs (Randomized) From Individualized Regimen(cPSS > 2)
Number analyzed (Participants) | 26 | 19
participants | 3 | 2

14. Secondary Outcome: Change in Fasting Non-HDL Cholesterol From Baseline
Description: Fasting non-HDL cholesterol calculated from difference between fasting total cholesterol and fasting HDL level. Missing values and non-fasting values excluded.
Time Frame: From study entry to Weeks 24, 48
Population: All randomized participants who started study treatment. Non-fasting results and missing results excluded from analysis. Therefore, differences reported here represent a complete case analysis.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Add NRTIs (Randomized) to Individualized Regimen (cPSS > 2.0) | Omit NRTIs (Randomized) From Individualized Regimen(cPSS > 2)
Number analyzed (Participants) | 180 | 177
mg/dL
  Change from baseline to week 24 (N=131; N=121) | 4.1 (35.8) | 20.8 (39.8)
  Change from baseline to week 48 (N=125 ; N=117) | 7.6 (35.5) | 19.8 (34.1)

15. Secondary Outcome: Participants With Newly Acquired HIV Drug Resistance Between Study Entry and Confirmed Virologic Failure
Description: Defined among the subgroup of participants experiencing the outcome of confirmed virologic failure. Newly acquired HIV drug resistance is defined as one or more ARVs with partial resistance or resistance when pre-entry resistance was fully sensitive or resistant when pre-entry resistance was fully sensitive or partially sensitive. The ARVs included for resistance acquisition included the following: darunavir/ritonavir; etravirine, tipranavir, tenofovir, emtracitabine, lamivudine, zidovudine, abacavir.
Time Frame: Between baseline and confirmed virologic failure (up to 96 weeks)
Population: Those with confirmed virologic failure (N=54; N=50) among the randomized arms included; and those who were missing resistance information following virologic failure (N=2; N=4) are excluded.
Measure: Number; unit: participants
Arm/Group | Add NRTIs (Randomized) to Individualized Regimen (cPSS > 2.0) | Omit NRTIs (Randomized) From Individualized Regimen(cPSS > 2)
Number analyzed (Participants) | 52 | 46
participants | 18 | 13

ADVERSE EVENTS:
Time Frame: AE data collected between date of first dose of study Rx, and end of week 96 study visit window (up to 110 weeks post entry), which may include follow-up/events after PCD . Those who never started study Rx are excluded from AE evaluation and analysis.
Description: Randomized arms only. All SAEs (per ICH, regardless of relationship to treatment), all cancers, MIs and hepatic failures; grade>2 signs/symptoms per ACTG criteria; all AST, ALT, creatinine, creatinine clearance, urinalysis, fasting lipid & glucose, and other Grade>2 labs, and all S/Sx or labs that lead to a change in study treatment were requested.
Groups:
- Omit NRTIs (Randomized) to Individualized Regimen (cPSS > 2.0): Individualized ARV study regimen with antiretroviral potency defined as continuous phenotype sensitivity score (cPSS) greater than 2.0 recommended and chosen prior to randomization. To this regimen, an individualized NRTI combination of at least 2 drugs from this class, chosen prior to randomization, was omitted, and any NRTIs the participant had been taking prior to randomization were to be permanently discontinued.
Arm/Group | Add NRTIs (Randomized) to Individualized Regimen (cPSS > 2.0) | Omit NRTIs (Randomized) to Individualized Regimen (cPSS > 2.0)
Serious Adverse Events (participants affected / at risk) | 58/180 | 49/177
Other Adverse Events (participants affected / at risk) | 169/180 | 165/177
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Add NRTIs (Randomized) to Individualized Regimen (cPSS > 2.0) (N=180) | Omit NRTIs (Randomized) to Individualized Regimen (cPSS > 2.0) (N=177)
Anaemia (Blood and lymphatic system disorders) | 2 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 2
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 1
Angina unstable (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 2
Hyperthyroidism (Endocrine disorders) | 1 | 0
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Ascites (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Intestinal fistula (Gastrointestinal disorders) | 0 | 1
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1
Chest pain (General disorders) | 6 | 6
Death (General disorders) | 0 | 1
Device dislocation (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 2
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Hepatotoxicity (Hepatobiliary disorders) | 1 | 0
Autoimmune disorder (Immune system disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 2
Immune reconstitution inflammatory syndrome (Immune system disorders) | 1 | 0
AIDS dementia complex (Infections and infestations) | 1 | 0
Abdominal wall infection (Infections and infestations) | 0 | 1
Abscess of salivary gland (Infections and infestations) | 0 | 1
Acute hepatitis B (Infections and infestations) | 0 | 1
Arthritis bacterial (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1
Bronchopneumonia (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 4
Diverticulitis (Infections and infestations) | 0 | 1
Endometritis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 3
Gastroenteritis viral (Infections and infestations) | 0 | 1
Genital herpes (Infections and infestations) | 1 | 0
HIV wasting syndrome (Infections and infestations) | 1 | 0
Herpes oesophagitis (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 2
Influenza (Infections and infestations) | 0 | 1
Laryngitis (Infections and infestations) | 1 | 0
Liver abscess (Infections and infestations) | 0 | 1
Lobar pneumonia (Infections and infestations) | 1 | 1
Meningitis listeria (Infections and infestations) | 1 | 0
Mycobacterium avium complex infection (Infections and infestations) | 0 | 1
Parvovirus infection (Infections and infestations) | 1 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 7 | 6
Pneumonia bacterial (Infections and infestations) | 2 | 2
Pneumonia viral (Infections and infestations) | 1 | 0
Post procedural infection (Infections and infestations) | 1 | 0
Postoperative wound infection (Infections and infestations) | 0 | 1
Progressive multifocal leukoencephalopathy (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 0 | 3
Urinary tract infection (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 2 | 1
Gun shot wound (Injury, poisoning and procedural complications) | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Multiple fractures (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Hepatic enzyme increased (Investigations) | 0 | 1
Transaminases increased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Gout (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0
Adenosquamous cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 2
Convulsion (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Neurological symptom (Nervous system disorders) | 0 | 1
Radiculopathy (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 1
VIIth nerve paralysis (Nervous system disorders) | 1 | 1
Bipolar I disorder (Psychiatric disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 1
Mood altered (Psychiatric disorders) | 0 | 1
Substance abuse (Psychiatric disorders) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 1 | 2
Suicide attempt (Psychiatric disorders) | 1 | 2
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1
Testicular torsion (Reproductive system and breast disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Physical assault (Social circumstances) | 0 | 1
Bartholin's cyst removal (Surgical and medical procedures) | 0 | 1
Colostomy (Surgical and medical procedures) | 0 | 1
Finger amputation (Surgical and medical procedures) | 1 | 0
Inguinal hernia repair (Surgical and medical procedures) | 1 | 0
Intervertebral disc operation (Surgical and medical procedures) | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1
Venous thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Add NRTIs (Randomized) to Individualized Regimen (cPSS > 2.0) (N=180) | Omit NRTIs (Randomized) to Individualized Regimen (cPSS > 2.0) (N=177)
Diarrhoea (Gastrointestinal disorders) | 8 | 9
Nausea (Gastrointestinal disorders) | 12 | 6
Fatigue (General disorders) | 9 | 8
Pyrexia (General disorders) | 7 | 11
Bronchitis (Infections and infestations) | 12 | 12
Herpes simplex (Infections and infestations) | 6 | 9
Herpes zoster (Infections and infestations) | 5 | 10
Oral candidiasis (Infections and infestations) | 10 | 6
Pneumonia bacterial (Infections and infestations) | 12 | 11
Upper respiratory tract infection (Infections and infestations) | 16 | 14
Urinary tract infection (Infections and infestations) | 4 | 9
Alanine aminotransferase increased (Investigations) | 38 | 41
Aspartate aminotransferase increased (Investigations) | 50 | 47
Blood alkaline phosphatase increased (Investigations) | 11 | 4
Blood bilirubin increased (Investigations) | 9 | 6
Blood cholesterol (Investigations) | 8 | 11
Blood cholesterol abnormal (Investigations) | 70 | 82
Blood cholesterol increased (Investigations) | 11 | 22
Blood creatinine increased (Investigations) | 26 | 30
Blood glucose abnormal (Investigations) | 54 | 62
Blood glucose decreased (Investigations) | 19 | 15
Blood glucose increased (Investigations) | 30 | 37
Blood potassium decreased (Investigations) | 3 | 9
Blood triglycerides (Investigations) | 12 | 12
Low density lipoprotein (Investigations) | 17 | 22
Low density lipoprotein abnormal (Investigations) | 48 | 47
Low density lipoprotein increased (Investigations) | 9 | 13
Neutrophil count decreased (Investigations) | 21 | 9
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 | 6
Headache (Nervous system disorders) | 14 | 13
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12 | 3
Hypertension (Vascular disorders) | 6 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In accordance with the Clinical Trials Agreement between NIAID (DAIDS) and company collaborators, NIAID (DAIDS) provides companies with a copy of any abstract, press release, or manuscript prior to submission for publication with sufficient time for company review and comment. The publication/other disclosure can be delayed for up to 30 additional business days for manuscripts and five (5) business days for abstracts, to preserve U.S. or foreign patent or other intellectual property rights.